CLINICAL TRIAL: NCT03200990
Title: PULsecath mechanicaL Support Evaluation (PULSE) - Trial
Brief Title: PULsecath mechanicaL Support Evaluation
Acronym: PULSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, MD,PhD, Cardiologist, Principal Investigator, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pulse version 2.9
Record Dates: First submitted 2017-06-08; First posted 2017-06-28 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease; Heart Failure; Cardiogenic Shock
Keywords: pressure-volume loops; cardiac mechanics; high-risk PCI
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- iVAC2L pVAD (Experimental): Clinically indicated ventricular support for high-risk PCI with Pulsecath iVAC2L.
  Interventions: Device: iVAC2L pVAD

INTERVENTIONS:
Device: iVAC2L pVAD — To determine the effects of the new PFLVAD PulseCath® iVAC2L on ventricular loading using left ventricular pressure-volume loops, in association with systemic and pulmonary hemodynamic parameters obtained from right and left catheterization. Additionally, assessments of specific load and flow-dependent humoral factors, and cardiac enzymes, will be made during and after the use of mechanical circulatory support.

SUMMARY:
The objective of this study is to determine ventricular loading conditions during and after PulseCath® iVAC2L support, and assess its impact on specific load dependent humoral factors and cardiac enzymes. These specific patterns are so far unknown and will be evaluated invasively.

DETAILED DESCRIPTION:
This is a mechanistic exploratory study. The objective is to determine the effects of the new PFLVAD PulseCath® iVAC2L on ventricular loading using left ventricular pressure-volume loops, in association with systemic and pulmonary hemodynamic parameters obtained from right and left catheterization. Additionally, assessments of specific load and flow-dependent humoral factors and cardiac enzymes will be made during and after the use of mechanical circulatory support. These specific patterns are so far unknown. Knowledge of optimal patterns may help in determining the ideal circulatory device platform.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥ 18 years;
2. Informed Consent must be signed by the patient, prior to HR-PCI;
3. The multidisciplinary heart team has reached consensus for high-risk PCI. Patients may present with left ventricular systolic dysfunction (ejection fraction ≤40%);
4. Anatomical criteria: Intervention to an unprotected left main coronary artery, left main equivalent or single remaining vessel; multivessel disease; intervention in a distal left main bifurcation.

Exclusion Criteria:

1. No written informed consent;
2. Left ventricular thrombus;
3. Interventricular septal defect;
4. Significant peripheral arterial disease or arterial lumen size < 6mm at the level of the common femoral artery;
5. Significant aortic valve disease (more than mild aortic stenosis/regurgitation);
6. Cardiogenic shock;
7. Previous stroke within the last 3 months;
8. Major bleeding event within last 3 months;
9. Chronic kidney disease with a GFR < 25 mL/min;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pressure-volume Area (PVA) | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Myocardial Oxygen Consumption (MVO2) following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in PVA will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg.mL

SECONDARY OUTCOMES:
Change in Cardiac Output | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Cardiac Output (CO), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in CO will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: L/min
Change on the Mean Pulmonary Capillary Wedge Pressure | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Mean Pulmonary Capillary Wedge Pressure (mPCWP), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in mPCWP will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg.
Change in the PCWP v-wave | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in PCWP v-wave (vPCWP), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in vPCWP will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg.
Change in Mean Pulmonary Artery Pressure | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Mean Pulmonary Artery Pressure (mPAP), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in mPAP will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg.
Change in Pulmonary Artery Oxygen Saturation | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Pulmonary Artery Oxygen Saturation, also known as Mixed Oxygen Saturation (SVO2), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in SVO2 will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: %
Change in Right Atrial Pressure | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Right Atrial Pressure (RAP), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in RAP will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg.
Change in Preload-recruitable Stroke Work | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in Preload-recruitable Stroke Work (PRSW), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in PRSW will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg
Change in the Starling Contractile Index | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in the Starling Contractile Index (SCI), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in SCI will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg/ml⋅s
Change in End-systolic Wall Stress | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in the End-systolic Wall Stress (WSes), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in WSes will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg.
Change in the first derivative of pressure over time | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in the first derivative of pressure over time (+dP/dtmax), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in +dP/dtmax will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: mmHg/s
Change in Systemic Vascular Resistance | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in the Systemic Vascular Resistance (SVR), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in SVR will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: (dyn∙s)/(cm^(-5))
Change in Pulmonary Vascular Resistance | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in the Pulmonary Vascular Resistance (PVR), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in PVR will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: (dyn∙s)/(cm^(-5))
Change in Cardiac Power Output | From the beginning of the PCI until its conclusion. This period can be variable and is estimated in 40 to 270 minutes.
  Numerical continuous variable representing the change in the Cardiac Power Output (CPO), following ventricular unloading. The PULSE trial will measure in real-time how discrepant this measurement can be when resulting from continuous or pulsatile flow ventricular assist devices. This is not a time-to-event outcome: the change in CPO will be obtained from real-time data collected during the intervention. The time frame will be the time of the Intervention. Unit: Watts
Change in Hematocrit | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in Hematocrit (Ht) as an indicative of bleeding or hemolysis. Unit: %
Change in Hemoglobin | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in Hemoglobin (Hb) as an indicative of bleeding or hemolysis. Unit: mmol/L
Change in Platelet Count | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in Platelet Count as an indicative of bleeding events. Unit: 10^9/L
Change in haptoglobin | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in haptoglobin as an indicative of hemolytic events. Unit: g/L
Change in total and conjugated bilirubin | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in total and conjugated bilirubin as an indicative of hemolytic events. Unit: umol/L
Change in lactate dehydrogenase | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in lactate dehydrogenase as an indicative of hemolytic events. Unit: U/L.
Change in hs-troponin | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in hs-troponin as an indicative of myocardial necrosis. Unit: ng/L
Change in creatinephosphokinase | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in creatinephosphokinase (CK) as an indicative of myocardial necrosis. Unit: U/L
Change in creatinophosphokinase MB mass assay | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in creatinophosphokinase MB mass assay (CKMB-mass) as an indicative of myocardial necrosis. Unit: ug/L
Change in N-terminal pro b-type natriuretic peptide | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in N-terminal pro b-type natriuretic peptide (NT-proBNP) as an indicative of chamber overload. Unit: pmol/L
Change in serum lactate | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in serum lactate as an indicative of hypoperfusion states. Unit: mmol/L.
Change in serum creatinine | From baseline (beginning of PCI) to immediately after the procedure and 12 hours after PCI.
  Numerical continuous variable. Change in serum creatinine as an indicative of acute kidney injury. Unit: umol/L
All-cause mortality | 30 days follow up
  Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG). Time-to-event variable, measured in days.
Acute myocardial infarction | 30 days follow up
  According to the "Fourth Universal Definition of Acute Myocardial Infarction". Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG). Time-to-event variable, measured in days.
Stroke or transient ischemic attack | 30 days follow up
  As per VARC 2 definitions 2013 J Thorac Cardiovasc Surg 2013;145:6-23. Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG). Time-to-event variable, measured in days.
Repeat revascularization | 30 days follow up
  As per ARC definition - Circulation. 2007;115:2344-2351. Constitutes one of the components of the MACCE composite endpoint: all-cause mortality, acute myocardial infarction, stroke or transient ischemic attack (TIA), and repeat revascularization (PCI or CABG). Time-to-event variable, measured in days.
Major Bleeding | 30 days follow up
  Major bleeding (BARC 3 to 5), according to the BARC Bleeding Classification (BARC definitions 2011. Circulation. 2011; 123(23): 2736-47. Time-to-event variable, measured in days.
Major vascular complications | 30 days follow up
  Major vascular complications (e.g.: arteriovenous fistula, limb ischemia), as per VARC-2 definitions (VARC 2 definitions 2013, J Thorac Cardiovasc Surg 2013;145:6-23) . Time-to-event variable, measured in days.
Acute renal dysfunction | 30 days follow up
  Acute renal dysfunction (AKIN 1 or above), using the AKIN Classification as described in the VARC-2 definitions (VARC 2 definitions 2013 J Thorac Cardiovasc Surg 2013;145:6-23).
Increase in Aortic regurgitation | 30 days follow up
  Increase in aortic regurgitation by more than one grade (TTE). Binary outcome obtained at the second echocardiogram, performed at discharge.
Severe hypotension | First 48 hours after the start of PCI.
  Severe hypotension (MAP < 60mmHg for more than 10 minutes despite fluid resuscitation or use of vasoactive amines to maintain MAP ≥ 60 mm Hg), or shock, defined based on the definition from the SHOCK trial (1) SBP ≤ 90mmHg for at least 30 minutes, (2) Need for vasopressors to maintain SBP > 90mmHg; (3) evidence of end-organ hypoperfusion; (4) Evidence of elevated filling pressures. A similar concept has been applied in the BCIS-1 study to measure procedural instability (JAMA. 2010;304(8):867-874).
Ventricular arrhythmias | 30 days follow up
  VT requiring cardioversion and / or need for CPR. Binary outcome, VF at anytime during follow up. Time-to-event analysis, measured in days.
Angiographic failure | Assessed at the end of the PCI. This time point (end of PCI) can be variable and is estimated in 40 to 270 minutes after the beginning of the procedure.
  Angiographic failure/ procedural failure, as defined in the 2011 ACCF/AHA/SCAI Guideline for Percutaneous Coronary Intervention Circulation. 2011;124:e574-e651): post PCI TIMI flow < III, residual stenosis (>50% post-balloon or > 10% post stenting), or presence of thrombus, side branch loss or flow limiting dissection. It is a binary outcome (yes/no answer). No time-to-event analysis will be applied.
Time of hospitalization | 30 days follow up
  Time to hospital discharge (in days).
Change in Left ventricular ejection fraction | From baseline (beginning of PCI) to the moment of discharge, assessed up to 30 days.
  Numerical continuous variable. Change in LVEF measured by trans-thoracic echocardiography at baseline and discharge. Not a time-to-event variable. Unit: %

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas v. Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (3):
- Clinic Pasteur, Toulouse, France
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands
- Kings College London, St. Thomas' Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bastos MB, McConkey H, Malkin O, den Uil C, Daemen J, Patterson T, Wolff Q, Kardys I, Schreuder J, Lenzen M, Zijlstra F, Redwood S, Van Mieghem NM. Effect of Next Generation Pulsatile Mechanical Circulatory Support on Cardiac Mechanics: The PULSE Trial. Cardiovasc Revasc Med. 2022 Sep;42:133-142. doi: 10.1016/j.carrev.2022.03.013. Epub 2022 Mar 14. PMID 35331637
- [Derived] Dedic A, Bastos MB, Van Mieghem NM. Pressure-Volume Loop Analysis in Percutaneous Coronary Intervention-Induced Shock. JACC Case Rep. 2020 Sep 23;2(12):1882-1883. doi: 10.1016/j.jaccas.2020.07.026. eCollection 2020 Oct. PMID 34317072